CLINICAL TRIAL: NCT04365322
Title: Étude Des réponses Immunitaires Lymphocytaires spécifiques Chez Des Patients infectés Par le Virus SARS-CoV-2 : Caractéristiques Des Réponses Effectrices et Mémoires
Brief Title: Study of Specific Viral Immune Responses Induced by SARS-CoV-2 (COVID-19)
Acronym: COV-CREM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: 2020/502
Record Dates: First submitted 2020-04-25; First posted 2020-04-28 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-05

CONDITIONS: SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Severe COVID-19 infection
  Interventions: Other: Additional biological samples
- Light to moderate COVID-19 infection
  Interventions: Other: Additional biological samples
- Cancer patients with COVID-19 infection
  Interventions: Other: Additional biological samples

INTERVENTIONS:
Other: Additional biological samples — Peripheral Blood Mononuclear Cell (PBMC) and plasma will be collected.
  Other Names: Additional blood samples will be realized as part of the care

SUMMARY:
SARS-CoV-2, has caused an international outbreak of respiratory illness termed Covid-19. The investigators used peptides derived from SARS-CoV-2 virus, to study viral-specific immune responses. COV-CREM is a French prospective monocentric study that will evaluate viral-specific cell responses in positive patients for SARS-CoV-2 on the basis of (RT-PCR) assay performed in respiratory tract sample tested by our local Center for Disease Control.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 PCR positive,
* Hospitalized patients with illness of any duration, and/or SpO2 ≤ 92% on room air.
* Cohorte C : patients with cancer (hematological malignancies and solid tumors).

Exclusion Criteria:

* Refusal to participate,
* Any immunosuppressive therapy (i.e. corticosteroids >10mg of hydrocortisone or equivalent dose) within 14 days before the planned start of study,
* Active or chronic hepatitis B or C and/or HIV positive (HIV 1/2 antibodies patients), or a known history of active Tuberculosis bacillus,
* Active autoimmune disease that required a systemic treatment, with the following exceptions:

  * Patients with a history of autoimmune-related hypothyroidism who are on thyroid replacement hormone are eligible for the study,
  * Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study,
* Prior allogeneic bone marrow transplantation or prior solid organ transplantation,
* Patients currently exposed to chemotherapy, anti-tumor immunotherapy as anti-PD-1, anti-PD-L1, or anti-CTLA4 agent or any immune therapy or biotherapy (except for patients in cohort C),
* Previous prescribing of biotherapy or treatment for the management of COVID-19 is not an exclusion criterion,
* Patient under guardianship, curatorship or under the protection of justice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with COVID-19 or convalescent.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2020-04-20 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2025-04-20 (Estimated)

PRIMARY OUTCOMES:
Specific immune responses | During COVID-19 infection or one month after COVID-19 infection
  Intensity and diversity of immune responses specific for SARS-COV-2

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Jean Minjoz, Besançon, France